CLINICAL TRIAL: NCT01448707
Title: PROTEAse Inhibitor (DRV/Rtv) in Mono- or Triple Therapy in Suppressed HIV-1 Infected Subjects
Brief Title: A Clinical Trial Comparing the Efficacy of Darunavir/Ritonavir Monotherapy Versus a Triple Combination Therapy Containing Darunavir/Ritonavir and 2 Nucleoside/Nucleotide Reverse Transcriptase Inhibitors in Patients With Undetectable Plasma HIV-1 RNA on Current Treatment
Acronym: PROTEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR018370; TMC114IFD3003 (Other: Janssen); 2011-001635-23 (EudraCT Number); PROTEA (Other: Janssen)
Record Dates: First submitted 2011-06-02; First posted 2011-10-07 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-10

CONDITIONS: Human Immunodeficiency Virus (HIV) Infections; Acquired Immunodeficiency Syndrome (AIDS) Virus
Keywords: Darunavir (DRV); TMC114; Prezista; HIV; virologic response; neurocognitive function
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections; Virus Diseases | interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Darunavir monotherapy (Experimental): Darunavir (DRV) + ritonavir (rtv): 2 tablets DRV 400 mg should be taken together with 1 tablet rtv 100 mg within 30 minutes after a meal. Following the primary efficacy analysis after Week 48, patients who entered the study with a nadir CD4+ count of <200 cells/μL will also receive 2 N[t]RTIs (ie, triple therapy) as soon as possible
  Interventions: Drug: Darunavir; Drug: Ritonavir
- Triple therapy containing darunavir (Active Comparator): Darunavir (DRV) + ritonavir (rtv) + 2 N[t]RTIs: 2 tablets DRV 400 mg should be taken together with 1 tablet rtv 100 mg within 30 minutes after a meal in combination with 2 N[t]RTIs (an investigator-selected dual combination of either abacavir (ABC), lamivudine (3TC), zidovudine (AZT), tenofovir disoproxil fumarate (TDF) or emtricitabine (FTC)
  Interventions: Drug: Darunavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Darunavir — Darunavir (DRV): type = exact number, unit = mg, number = 800, form = tablet, route = oral use
Drug: Ritonavir — ritonavir (rtv): type = exact number, unit = mg, number = 100, form = tablet, route = oral use

SUMMARY:
The purpose of this study is to compare the efficacy, safety and tolerability of darunavir/ritonavir 800/100 mg monotherapy with a triple combination therapy containing darunavir/ritonavir 800/100 mg and 2 nucleoside/nucleotide reverse transcriptase inhibitors (N[t]RTIs) in approximately 260 Human Immunodeficiency Virus-1 (HIV-1) infected patients who have been on Highly Active AntiRetroviral Therapy (HAART) medication and have a plasma Viral Load below 50 copies/mL for at least 48 weeks. Also the changes in neurocognitive function will be compared throughout the study.

DETAILED DESCRIPTION:
This is phase IIIb, randomised (study medication is assigned by chance), open-label (both the patient and the study physician will know to which treatment group the patient is assigned) trial to compare the efficacy, safety and tolerability of darunavir/ritonavir (DRV/rtv) 800/100 mg once daily monotherapy with a triple combination therapy containing DRV/rtv 800/100 mg once daily and an investigator-selected background of 2 other anti-HIV drugs of the class nucleoside/nucleotide reverse transcriptase inhibitors (N[t]RTIs). The investigator-selected N[t]RTIs is a dual combination of either be abacavir (ABC), lamivudine (3TC), zidovudine (AZT), tenofovir disoproxil fumarate (TDF) or emtricitabine (FTC). Approximately 260 HIV-1 infected patients, who have received HAART for at least 48 weeks, have not changed their treatment within the last 8 weeks, and who have documented evidence of plasma viral load (plasma HIV-1 RNA) below 50 copies/mL for at least 48 weeks prior to being screened, participate in the study. The study period includes a screening period of maximum 6 weeks, a 4-week run-in period, a 96 week treatment period, followed by a 4 weeks follow-up period. According to the original protocol, at the start of the 4-week run-in period all patients replaced their 3rd agent (non-nucleoside reverse transcriptase (NNRTI), protease inhibitor (PI) or integrase inhibitor) of the HAART medication with DRV/rtv and continued with the 2 N[t]RTIs. After 4 weeks the patient was randomly assigned (like flipping a coin) to either the monotherapy group or the triple therapy group. If assigned to the monotherapy group, the 2 N[t]RTIs were stopped and only DRV/rtv was continued. If assigned to the triple therapy group, DRV/rtv were continued together with 2 N[t]RTIs, which can be the same as already taken or are switched to new N[t]RTIs. Based on the primary efficacy analysis after Week 48, the protocol was amended such that subjects in the monotherapy arm who entered the study with a nadir CD4+ count of <200 cells/μL will also receive 2 N[t]RTIs (ie, triple therapy) as soon as possible.

The main purpose of this study is to demonstrate that DRV/rtv monotherapy is as effective as a triple combination therapy containing DRV/rtv and 2N[t]RTIs. In addition, the study looks at overall safety and tolerability between the two treatment groups. During the study, patients' health are monitored by physical examination, checking of vital signs (blood pressure / pulse), and laboratory testing on blood and urine samples. Also blood samples are drawn to measure the antiviral effectiveness (i.e., decrease of the plasma viral load to a level <50 HIV-1 RNA copies/mL) and immunology assessments (to assess the body's immune system). A battery of neurocognitive function tests is performed during the study visits. A sub-study takes place in selected hospitals. Approximately 100 patients have 2 additional tests done, at the start of the run-in phase and after 48-weeks of randomisation. For this substudy a lumbar puncture (extraction of cerebrospinal fluid [CSF] from the spinal canal) for laboratory testing (antiviral effectiveness, pharmacokinetic analysis, biochemistry and immune markers) and an additional blood sample for pharmacokinetic analysis (to measure the drug level in blood) is taken. The study hypothesis is that, after 48 weeks of randomised treatment, DRV/rtv monotherapy is as effective as the triple therapy containing DRV/rtv plus 2 N[t]RTIs. Two 400 mg tablets of darunavir and one 100 mg tablet ritonavir are taken together once daily orally within 30 minutes after completion of a meal, for 100 weeks. The intake of the investigator-selected N[t]RTIs as according the local prescribing information.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* receiving HAART for at least 48 weeks
* Have at least 2 documented plasma HIV-1 RNA <50 copies/mL, and no HIV-1 RNA >=50 copies/mL in the 48 weeks prior to the screening
* Be taking the same antiretroviral (ARV) combination for at least 8 weeks before screening
* Have the preference, together with the physician, to change the current HAART regimen for reasons of simplification and/or toxicity

Exclusion Criteria:

* Has a history of virologic failure defined as 2 consecutive plasma HIV-1 RNA >500 copies/mL while on previous or current antiretroviral therapy
* Has a history of any primary PI mutations
* Has clinical or laboratory evidence of significantly decreased hepatic function or decompensation, irrespective of liver enzyme levels (liver insufficiency)
* Is diagnosed with acute viral hepatitis at screening or before Baseline 1
* Is co-infected with hepatitis B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2012-03-15 (Actual); Primary Completion 2014-06-11 (Actual); Study Completion 2015-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (34):
- Austria (2):
  - Graz
  - Vienna
- Belgium (3):
  - Antwerp
  - Brussels
  - Ghent
- Denmark (2):
  - Copenhagen
  - Hvidovre
- France (4):
  - Bobigny
  - Bondy
  - Dijon
  - Paris
- Germany (5):
  - Berlin
  - Bonn
  - Cologne
  - Frankfurt
  - Hanover
- Budapest, Hungary
- Ireland (2):
  - Dublin
  - Galway
- Israel (3):
  - Beersheba
  - Ramat Gan
  - Tel Aviv
- Warsaw, Poland
- Spain (5):
  - Badalona
  - Barcelona
  - Córdoba
  - Granada
  - Madrid
- Stockholm, Sweden
- Switzerland (2):
  - Sankt Gallen
  - Zurich
- United Kingdom (3):
  - Brighton
  - London
  - Manchester

REFERENCES:
- [Derived] Girard PM, Antinori A, Arribas JR, Ripamonti D, Bicer C, Netzle-Sveine B, Hadacek B, Moecklinghoff C. Week 96 efficacy and safety of darunavir/ritonavir monotherapy vs. darunavir/ritonavir with two nucleoside reverse transcriptase inhibitors in the PROTEA trial. HIV Med. 2017 Jan;18(1):5-12. doi: 10.1111/hiv.12386. Epub 2016 Jun 9. PMID 27279571

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 325 participants screened, among them 282 were eligible for run-in phase and among them 274 enrolled to the study. 1 randomized participant was not treated (274 participants were randomized).
Groups:
- DRV/Rtv MONO: Darunavir (DRV) and ritonavir (rtv): 2 tablets DRV 400 mg were taken together with 1 tablet rtv 100 mg within 30 minutes after a meal.
- DRV/Rtv + 2NRTIs: Darunavir (DRV), ritonavir (rtv) and 2 N[t]RTIs: 2 tablets DRV 400 mg were taken together with 1 tablet rtv 100 mg within 30 minutes after a meal in combination with 2 N[t]RTIs (an investigator-selected dual combination of either abacavir (ABC), lamivudine (3TC), zidovudine (AZT), tenofovir disoproxil fumarate (TDF) or emtricitabine (FTC).
Period: Overall Study
Arm/Group | DRV/Rtv MONO | DRV/Rtv + 2NRTIs
Started | 137 | 136
Completed | 119 | 118
Not Completed | 18 | 18
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 2 | 6
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Other | 7 | 4

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were analyzed for all participants who were treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | DRV/Rtv MONO | DRV/Rtv + 2NRTIs | Total
Number analyzed (Participants) | 137 | 136 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (11.21) | 43.1 (10.41) | 43.9 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 21 | 47
  Male | 111 | 115 | 226
Region of Enrollment [Number; unit: participants]
  AUSTRIA | 5 | 5 | 10
  BELGIUM | 7 | 8 | 15
  DENMARK | 8 | 7 | 15
  FRANCE | 16 | 12 | 28
  GERMANY | 11 | 11 | 22
  HUNGARY | 5 | 3 | 8
  IRELAND | 3 | 5 | 8
  ISRAEL | 5 | 5 | 10
  ITALY | 22 | 24 | 46
  POLAND | 7 | 6 | 13
  SPAIN | 17 | 23 | 40
  SWEDEN | 3 | 4 | 7
  SWITZERLAND | 10 | 5 | 15
  UNITED KINGDOM | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Virologic Response (Food Drug and Administration [FDA] Snapshot, Switch = Failure)
Description: The percentage of participants who have plasma human immunodeficiency virus type-1 (HIV-1) ribonucleic acid (RNA) levels <50 copies/milliliters [mL] after 48 weeks of follow-up. Switch = Failure is defined as switch in background nucleoside/nucleotide reverse transcriptase inhibitors (N[t]RTIs) not permitted by the trial protocol or plasma HIV-1 RNA assessment closest to target date of the analysis time point window (44-52 weeks) and next/confirmation of Plasma HIV-1 RNA in the analysis time point window above the threshold or discontinuation for any other reason.
Time Frame: Week 48
Population: The intent-to-treat (ITT) population is the set of all participants who were randomized and who took at least one dose of study medication in the treatment phase.
Measure: Number; unit: Percentage of Participants
Groups:
- DRV/r: Darunavir (DRV) + ritonavir (rtv): 2 tablets DRV 400 mg should be taken together with 1 tablet rtv 100 mg within 30 minutes after a meal.
- DRV/r + 2NRTIs: Darunavir (DRV) + ritonavir (rtv) + 2 N[t]RTIs: 2 tablets DRV 400 mg should be taken together with 1 tablet rtv 100 mg within 30 minutes after a meal in combination with 2 N[t]RTIs (an investigator-selected dual combination of either abacavir (ABC), lamivudine (3TC), zidovudine (AZT), tenofovir disoproxil fumarate (TDF) or emtricitabine (FTC)
Arm/Group | DRV/r | DRV/r + 2NRTIs
Number analyzed (Participants) | 137 | 136
Percentage of Participants | 87.0 | 95.0
Statistical Analysis 1: Comparison: DRV/r vs DRV/r + 2NRTIs; Test type: Non-Inferiority or Equivalence — Non-inferiority of DRV/rtv monotherapy versus triple therapy was assessed with a maximum allowable difference of 12 percent (%), with a one-sided significance level of 2.5%; p = 0.2331, Mixed Models Analysis — P-Value for non-inferiority of DRV/rtv MONO vs DRV/rtv + 2NRTIs (delta = 12%); Predicted response rate:confidence limits are obtained by means of logistic regression model with treatment group and Hepatitis C status as covariates; Non-Linear mixed = -7.9, 95% CI 2-sided [-14.64 to -1.19]

2. Secondary Outcome: Virologic Response (Food Drug and Administration [FDA] Snapshot, Switch = Failure)
Description: The percentage of participants who have plasma human immunodeficiency virus type-1 (HIV-1) ribonucleic acid (RNA) levels <50 copies/milliliters [mL] after 96 weeks of follow-up after switching to DRV/ritonavir(rtv) monotherapy versus triple therapy containing DRV/rtv. Switch = Failure is defined as switch in background nucleoside/nucleotide reverse transcriptase inhibitors (N[t]RTIs) not permitted by the trial protocol.
Time Frame: Week 96
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | DRV/r | DRV/r + 2NRTIs
Number analyzed (Participants) | 137 | 136
Percentage of Participants | 75.2 | 85.3
Statistical Analysis 1: Comparison: DRV/r vs DRV/r + 2NRTIs; Test type: Non-Inferiority or Equivalence — Non-inferiority of DRV/rtv monotherapy versus triple therapy was assessed with a maximum allowable difference of 12 percent (%), with a one-sided significance level of 2.5% and 80% power; p = 0.6933, Mixed Models Analysis; Non-Linear mixed = -10.1, 95% CI 2-sided [-19.50 to -0.73]

3. Secondary Outcome: Virologic Response (FDA Snapshot, Switch Included)
Description: The percentage of participants who have plasma human immunodeficiency virus type-1 (HIV-1) ribonucleic acid (RNA) levels <50 copies/milliliters [mL] after 48 and 96 weeks of follow-up after switching to DRV/ritonavir(rtv) monotherapy versus triple therapy containing DRV/rtv. Switch included is defined as all participants who discontinued randomized medication were followed up on their subsequent treatment.
Time Frame: Week 48 and 96
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | DRV/r | DRV/r + 2NRTIs
Number analyzed (Participants) | 137 | 136
Percentage of Participants
  Week 48 | 93.0 | 96.5
  Week 96 | 89.3 | 89.9
Statistical Analysis 1: Comparison: DRV/r vs DRV/r + 2NRTIs; Test type: Non-Inferiority or Equivalence — Week 48: Non-inferiority of DRV/rtv monotherapy versus triple therapy was assessed with a maximum allowable difference of 12 percent (%), with a one-sided significance level of 2.5% and 80% power; p = 0.0016, Mixed Models Analysis; Non-linear mixed model = -3.5, 95% CI 2-sided [-8.77 to 1.72]
Statistical Analysis 2: Comparison: DRV/r vs DRV/r + 2NRTIs; Test type: Non-Inferiority or Equivalence — Week 96: Non-inferiority of DRV/rtv monotherapy versus triple therapy was assessed with a maximum allowable difference of 12 percent (%), with a one-sided significance level of 2.5% and 80% power; p = 0.0022, Mixed Models Analysis; non-linear mixed model = -0.7, 95% CI 2-sided [-7.89 to 6.58]

4. Secondary Outcome: Change From Baseline in Global Neurocognitive Performance z-Score
Description: Change in neurocognitive function of DRV/rtv monotherapy versus triple therapy containing DRV/rtv over 48 and 96 weeks. Neurocognitive function will be measured by Hopkins Verbal Learning Test (verbal learning and memory), Colour Trail Test (psychomotor speed and cognitive flexibility) and Grooved Pegboard Test (psychomotor speed and fine motor function). Higher values for change in z-score represent an improvement in Neurocognitive Performance (NP).
Time Frame: Baseline, Week 48 and 96
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | DRV/r | DRV/r + 2NRTIs
Number analyzed (Participants) | 137 | 136
Units on a Scale
  Change at Week 48 | 0.39 (0.048) | 0.42 (0.057)
  Change at Week 96 | 0.63 (0.060) | 0.57 (0.057)

5. Secondary Outcome: Time to Loss of Virologic Response
Description: Time (in days) it takes to show loss of response per time to loss of virologic response (TLOVR) algorithm: confirmed HIV-1 RNA >= 50 copies/mL or premature discontinuation.
Time Frame: Baseline up to Week 96 or early withdrawal
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | DRV/r | DRV/r + 2NRTIs
Number analyzed (Participants) | 137 | 136
Days | NA (19.92) [NA to NA] — The event occurred in less than 50 percent of the participants. | NA (18.88) [NA to NA] — The event occurred in less than 50 percent of the participants.

6. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Phenotypic Drug Resistance
Description: The loss of treatment options of DRV/rtv monotherapy versus triple therapy containing DRV/rtv at Weeks 48 and 96, as defined by treatment-emergent phenotypic drug resistance. Drug resistance is classified as: 1) Confirmed HIV RNA >= 400 copies/mL, 2) Post-baseline phenotypic data and 3) Phenotypic resistance to any of the drug classes (NRTI, NNRTI, or PI).
Time Frame: At Weeks 48 and 96
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | DRV/r | DRV/r + 2NRTIs
Number analyzed (Participants) | 137 | 136
Participants
  Confirmed HIV RNA >= 400 copies/mL | 1 | 2
  Post-baseline phenotypic data | 2 | 1
  Phenotypic resistance to any of the drug classes | 0 | 0

7. Secondary Outcome: Number of Participants Reporting Resistance Mutations With Confirmed Virologic Failure Who Have HIV RNA >400 Copies/mL and Genotype Resistance Results
Description: The viral genotype of participants treated with DRV/rtv monotherapy versus triple therapy containing DRV/rtv over 48 and 96 weeks. Genotypic resistance (number of resistance mutations) at any time point when a participant had a confirmed plasma VL >400 copies/mL after randomization was performed per treatment group for the ITT population. Results were summarized based on individual treatment received: Darunavir resistance mutations, non-nucleoside reverse transcriptase inhibitor (NNRTI) mutations, nucleoside reverse transcriptase inhibitor (NRTI) mutations, protease inhibitor (PI) resistance mutations, PR mutations, RT mutations, extended NNRTI mutations, primary PI mutations.
Time Frame: Over 48 and 96 Weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | DRV/r | DRV/r + 2NRTIs
Number analyzed (Participants) | 137 | 136
Participants
  Participans with HIV RNA >= 400 copies/mL | 1 | 2
  Number of 0 Darunavir resistance mutations | 2 | 1
  Number of 0 NNRTI mutations | 2 | 0
  Number of 1 NNRTI mutations | 0 | 1
  Number of 1 PI resistance mutations | 1 | 0
  Number of 5 PI resistance mutations | 0 | 1
  Number of 6 PI resistance mutations | 1 | 0
  Number of 11 PR mutations | 0 | 1
  Number of 15 PR mutations | 1 | 0
  Number of 7 PR mutations | 1 | 0
  Number of 14 RT mutations | 1 | 0
  Number of 16 RT mutations | 0 | 1
  Number of 33 RT mutations | 1 | 0
  Number of extended 0 NNRTI mutations | 2 | 0
  Number of extended 1 NNRTI mutations | 0 | 1
  Number of primary 0 PI mutations | 2 | 1
  Number of participants with no mutations | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 96 weeks
Description: The Safety (SAF) population is the set of all participants who took at least one dose of study medication.
Arm/Group | DRV/Rtv MONO | DRV/Rtv + 2NRTIs
Serious Adverse Events (participants affected / at risk) | 18/137 | 14/136
Other Adverse Events (participants affected / at risk) | 61/137 | 47/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DRV/Rtv MONO (N=137) | DRV/Rtv + 2NRTIs (N=136)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Anal Fistula (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Tenderness (General disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cytomegalovirus Infection (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Groin Abscess (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 2 | 0
Meningitis (Infections and infestations) | 0 | 1
Pharyngitis Bacterial (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Shigella Infection (Infections and infestations) | 1 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Laryngeal Injury (Injury, poisoning and procedural complications) | 0 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Anogenital Warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central Nervous System Lesion (Nervous system disorders) | 0 | 1
Encephalomyelitis (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Optic Neuritis (Nervous system disorders) | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Alcoholism (Psychiatric disorders) | 1 | 0
Substance Abuse (Psychiatric disorders) | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Excessive Granulation Tissue (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Gastrectomy (Surgical and medical procedures) | 0 | 1
Tonsillectomy (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DRV/Rtv MONO (N=137) | DRV/Rtv + 2NRTIs (N=136)
Diarrhoea (Gastrointestinal disorders) | 18 | 10
Fatigue (General disorders) | 7 | 7
Pyrexia (General disorders) | 4 | 7
Nasopharyngitis (Infections and infestations) | 16 | 11
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 4
Headache (Nervous system disorders) | 8 | 9
Depression (Psychiatric disorders) | 4 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Rash (Skin and subcutaneous tissue disorders) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days. The sponsor will not mandate modifications to scientific content and does not have the right to suppress information.